CLINICAL TRIAL: NCT02520544
Title: THE ATX REGISTRY ATX Register Accolade Stem & Trident/Tritanium Cup With X3 Insert International Multicentre Surveillance Register
Brief Title: ATX Register Accolade Stem & Trident/Tritanium Cup With X3 Insert
Acronym: ATX
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H-S-038
Record Dates: First submitted 2015-06-11; First posted 2015-08-13 (Estimated); Results first posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-10

CONDITIONS: Arthroplasty, Replacement, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Accolade stem (Active Comparator): All patients in a participating centre matching all of the inclusion criteria and none of the exclusion criteria and who receive the Accolade or Accolade II stem and Trident/Tritanium cup with X3 liner.
  Interventions: Device: Accolade stem; Device: Trident/Tritanium cup
- Accolade II stem (Active Comparator): All patients in a participating centre matching all of the inclusion criteria and none of the exclusion criteria and who receive the Accolade or Accolade II stem and Trident/Tritanium cup with X3 liner.
  Interventions: Device: Accolade II stem; Device: Trident/Tritanium cup

INTERVENTIONS:
Device: Accolade stem — Total hip replacement
  Arms: Accolade stem
Device: Accolade II stem — Total hip replacement
  Arms: Accolade II stem
Device: Trident/Tritanium cup — Total hip replacement

SUMMARY:
The aim of this register is to determine the Accolade/Accolade II stem and Trident/Tritanium cup survivorship over years.

DETAILED DESCRIPTION:
This is a prospective international multicentre surveillance register. The aim of this register is to determine the Accolade/Accolade II stem and Trident/Tritanium cup survivorship over years. All institutions willing to participate to the register, able to recruit at least 20 patients (up to 100 patients)

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female patients between 18-75 years of age.
2. Patients requiring uncemented primary Total Hip Arthroplasty (THA), suitable for the use of the Accolade stem and Trident/Tritanium cup.
3. Patients with a diagnosis of osteoarthritis (OA).
4. Patients who understand the conditions of the study and are willing and able to comply with the post-operative scheduled clinical and radiographic evaluations and the prescribed rehabilitation.
5. Patients who signed the Ethics Committee approved Informed Consent Form prior to surgery.

Exclusion Criteria:

1. Patients who require revision of a previously implanted hip prosthesis.
2. Patients who had a THA on contralateral side within the last 6 months.
3. Patients who had a THA on contralateral side more than 6 months ago and the rehabilitation period outcome was considered unsatisfactory or not good (Harris Hip Score < 85).
4. Patients who will need lower limb joint replacement for another joint within one year.
5. Patients requiring bilateral hip replacement.
6. Patients who have had a prior procedure of acetabular osteotomy.
7. Patients with acute femoral fractures
8. Obese patients where obesity is severe enough to affect subject's ability to perform activities of daily living (body mass index, kg/m2: BMI ≥ 35).
9. Patients with active or suspected infection.
10. Patients with malignancy - active malignancy.
11. Patients with severe osteoporosis, rheumatoid arthritis (RA), Paget's disease or renal osteodystrophy.
12. Patients immunologically suppressed, or receiving steroids in excess of physiologic dose requirements.
13. The patient has a neuromuscular or neurosensory deficit which would limit the ability to assess the performance of the device or the patient has a neurological deficit which interferes with the patient's ability to limit weight bearing or places an extreme load on the implant during the healing period.
14. Female patients planning a pregnancy during the course of the study.
15. Patients with systemic or metabolic disorders leading to progressive bone deterioration.
16. Patients, who as judged by the surgeon, are mentally incompetent or are unlikely to be compliant with the prescribed post-operative routine and follow-up evaluation schedule.
17. Patients with other severe concurrent joint involvements, which can affect their outcome.
18. Patients with other concurrent illnesses, which are likely to affect their outcome such as sickle cell anaemia, systemic lupus erythematosus or renal disease requiring dialysis.
19. Patient with a known sensitivity to device materials.
20. Patients under the protection of law (e.g. guardianship).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 472 (Actual)
Dates: Start 2012-01; Primary Completion 2024-11-12 (Actual); Study Completion 2024-11-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Bolder, MD, Principal Investigator — Amphia Zieknhuis Breda
Locations (8):
- Ziekenhuis Netwerk Antwerpen, Antwerp, Belgium
- Netherlands (5):
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - Amphia Ziekenhuis, Breda
  - Maatschap Orthopaedie Ikazia, Rotterdam
  - Orbis Medisch Concern, Sittard
  - Rijnstate Arnhem, Zevenaar
- Skånevård Kryh Division Kirurgi och Ortopedkliniken Hässleholm, Hässleholm, Sweden
- Harrogate and District NHS Foundation Trust, Harrogate, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 472 participants that were enrolled into the study between January 2012 and February 2015.
Pre-assignment Details: Of the 472 participants enrolled, 49 cases were censored and excluded from the final analysis. 23 cases did not have a study device implanted, 4 cases did not have their surgery performed, 1 case voluntarily withdrew, 1 case had surgery performed after enrolment window, and 20 cases had inclusion/exclusion criteria violations. Of the remaining 423 participants, there were no bilateral cases.
Period: Overall Study
Arm/Group | Accolade Stem | Accolade II Stem
Started | 289 | 134
Completed | 229 | 102
Not Completed | 60 | 32
Not completed — Death | 18 | 8
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrawal by Subject | 23 | 11
Not completed — Revision/Removal of Study Device | 11 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Accolade Stem | Accolade II Stem | Total
Number analyzed (Participants) | 289 | 134 | 423
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.71 (7.46) | 59.76 (8.01) | 60.41 (7.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 161 | 72 | 233
  Male | 128 | 62 | 190
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Netherlands | 267 | 45 | 312
  Sweden | 0 | 32 | 32
  Belgium | 22 | 24 | 46
  United Kingdom | 0 | 33 | 33

OUTCOME MEASURES:

1. Primary Outcome: Survivorship of the Device
Description: Survivorship shown in Kaplan Meier survival curves (statistic used to estimate the survival function from lifetime data).
Time Frame: 10 years Follow-up
Population: Outcome value for the 10-year post-operative timepoint is provided.
Measure: Number (95% Confidence Interval); unit: percentage of participants not revised
Arm/Group | Accolade Stem | Accolade II Stem
Number analyzed (Participants) | 289 | 134
percentage of participants not revised | 97.03 [94.15 to 98.51] | 98.27 [93.19 to 99.57]
Statistical Analysis 1: Comparison: Accolade Stem vs Accolade II Stem; Test type: Superiority; p = 0.4551, Log Rank

2. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With Modified Harris Hip Score (HHS) Patient Questionnaire
Description: Scores can range from 0 to 100 with 0 being the worst and 100 being the best score. A score of 80-100 is considered good-excellent and a score of less than or equal to 79 is considered fair-poor. 90-100 = excellent 80-89 = good 70-79 = fair 0-69 = poor
Time Frame: pre-operative, 1, 3, 5, 7 and 10 years follow-up
Population: Outcome values for the modified HHS provided at pre-operative and all post-operative timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Accolade Stem | Accolade II Stem
Number analyzed (Participants) | 289 | 134
units on a scale
  Preoperative: number analyzed (Participants) | 289 | 133
  Preoperative | 59.73 (11.60) | 58.47 (11.08)
  1 year: number analyzed (Participants) | 270 | 126
  1 year | 95.08 (8.58) | 93.34 (9.61)
  3 years: number analyzed (Participants) | 231 | 118
  3 years | 94.89 (8.10) | 95.07 (7.69)
  5 years: number analyzed (Participants) | 230 | 107
  5 years | 95.37 (8.32) | 95.39 (8.10)
  7 years: number analyzed (Participants) | 219 | 102
  7 years | 94.08 (9.19) | 94.24 (8.93)
  10 years: number analyzed (Participants) | 216 | 102
  10 years | 93.73 (9.77) | 94.23 (9.20)

3. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With Oxford Hip Score Patient Questionnaire
Description: Outcome instrument which contains 12 questions on activities of daily living that assess function and residual pain in patients undergoing total hip replacement (THR) surgery, each scored from 0-4 (worst to best), giving a final score with a total range of 0-48. A final score of 0 to 19 indicates severe hip arthritis, 20-29 indicates moderate to severe symptoms, 30-39 indicates mild to moderate symptoms, and 40 to 48 indicates satisfactory joint function.
Time Frame: pre-operative, 1, 3, 5, 7 and 10 years follow-up
Population: OHS values provided for pre-operative and all post-operative follow up timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Accolade Stem | Accolade II Stem
Number analyzed (Participants) | 289 | 134
units on a scale
  Pre-operative: number analyzed (Participants) | 289 | 130
  Pre-operative | 24.55 (8.06) | 22.47 (7.54)
  1 year: number analyzed (Participants) | 266 | 120
  1 year | 43.98 (5.60) | 44.20 (5.25)
  3 years: number analyzed (Participants) | 231 | 121
  3 years | 44.70 (5.36) | 44.84 (4.72)
  5 years: number analyzed (Participants) | 232 | 106
  5 years | 45.16 (5.23) | 45.79 (3.82)
  7 years: number analyzed (Participants) | 221 | 103
  7 years | 45.14 (4.97) | 44.49 (5.91)
  10 years: number analyzed (Participants) | 229 | 99
  10 years | 44.98 (4.66) | 44.75 (5.05)

4. Secondary Outcome: Investigation of Clinical Performance and Patient Outcome With EuroQuol-5 Dimension (EQ-5D) Patient Questionnaire
Description: The EQ-5D is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas: the EQ visual analogue scale (EQ VAS) and the EQ-5D descriptive system, time trade-off (TTO).
  The EQ VAS collects health state values using a 20 cm visual analogue scale with the endpoints labeled best imaginable health state at the top and worst imaginable health state at the bottom, having numeric values of 100 to 0 respectively.
  The EQ-5D Time Trade-off (TTO) descriptive system comprises the following five dimensions: mobility, self-care, usual activities, pain/comfort and anxiety/depression. Each dimension has three levels: no problems, some problems and extreme problems. The TTO index values on a scale between -1(low) and 1(high) show the average health status according to the 5 dimensions. A low score shows worse health, and a high score shows better health.
Time Frame: pre-operative, 1, 3, 5, 7 and 10 years follow-up
Population: EQ-5D values are provided for the VAS and TTO scores at the preoperative and all postoperative follow up timepoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Accolade Stem | Accolade II Stem
Number analyzed (Participants) | 289 | 134
units on a scale
  EQ-5D VAS Preoperative: number analyzed (Participants) | 289 | 130
  EQ-5D VAS Preoperative | 66.8 (16.9) | 66.9 (19.0)
  EQ-5D VAS 1 year follow up: number analyzed (Participants) | 263 | 119
  EQ-5D VAS 1 year follow up | 81.3 (12.4) | 83.1 (14.8)
  EQ-5D VAS 3 years follow up: number analyzed (Participants) | 230 | 121
  EQ-5D VAS 3 years follow up | 79.7 (13.1) | 81.0 (14.5)
  EQ-5D VAS 5 years follow up: number analyzed (Participants) | 231 | 106
  EQ-5D VAS 5 years follow up | 79.8 (14.2) | 81.1 (15.3)
  EQ-5D VAS 7 years follow up: number analyzed (Participants) | 220 | 102
  EQ-5D VAS 7 years follow up | 78.3 (14.2) | 79.6 (15.2)
  EQ-5D VAS 10 years follow up: number analyzed (Participants) | 222 | 102
  EQ-5D VAS 10 years follow up | 77.7 (14.3) | 78.2 (13.8)
  EQ-5D TTO Preoperative: number analyzed (Participants) | 289 | 130
  EQ-5D TTO Preoperative | 0.505 (0.260) | 0.471 (0.284)
  EQ-5D TTO 1 year follow up: number analyzed (Participants) | 265 | 119
  EQ-5D TTO 1 year follow up | 0.871 (0.185) | 0.866 (0.201)
  EQ-5D TTO 3 years follow up: number analyzed (Participants) | 231 | 121
  EQ-5D TTO 3 years follow up | 0.874 (0.185) | 0.846 (0.218)
  EQ-5D TTO 5 years follow up: number analyzed (Participants) | 231 | 107
  EQ-5D TTO 5 years follow up | 0.865 (0.210) | 0.891 (0.180)
  EQ-5D TTO 7 years follow up: number analyzed (Participants) | 222 | 103
  EQ-5D TTO 7 years follow up | 0.849 (0.201) | 0.866 (0.213)
  EQ-5D TTO 10 years follow up: number analyzed (Participants) | 224 | 102
  EQ-5D TTO 10 years follow up | 0.846 (0.227) | 0.867 (0.195)

ADVERSE EVENTS:
Time Frame: The study period during which AEs must be reported is defined as the period from the initiation of any study procedures to end of the study treatment follow-up. The start of study procedures is considered to be the date of consent. Adverse events were collected pre-operatively after enrolment and prior to surgery, intra-operatively, and over the 10-year post-operative time period up until the point of study termination.
Arm/Group | Accolade Stem | Accolade II Stem
All-Cause Mortality (participants affected / at risk) | 18/289 | 8/134
Serious Adverse Events (participants affected / at risk) | 92/289 | 56/134
Other Adverse Events (participants affected / at risk) | 36/289 | 41/134
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Accolade Stem (N=289) | Accolade II Stem (N=134)
Acetabular Insert Crack / Fracture - Operative Site (Musculoskeletal and connective tissue disorders) | 1 | 0
Dislocation - Operative Site (Musculoskeletal and connective tissue disorders) | 3 | 4
Excessive Hip Pain - Operative Site (Musculoskeletal and connective tissue disorders) | 1 | 0
Femoral Component Loosening - Operative Site (Musculoskeletal and connective tissue disorders) | 5 | 0
Femoral Component Subsidence - Operative Site (Surgical and medical procedures) | 1 | 0
Femoral Crack / Fracture - Operative Site (Musculoskeletal and connective tissue disorders) | 1 | 1
Superficial Wound Infection - Operative Site (Infections and infestations) | 2 | 0
Superficial Wound Infection - Operative Site (Skin and subcutaneous tissue disorders) | 0 | 1
Tendonitis - Operative Site (Musculoskeletal and connective tissue disorders) | 1 | 0
Wound Hematoma - Operative Site (Injury, poisoning and procedural complications) | 3 | 0
Wound Related - Operative Site (Infections and infestations) | 1 | 1
Wound Related - Operative Site (Skin and subcutaneous tissue disorders) | 2 | 0
Osteolysis - Operative Site (Musculoskeletal and connective tissue disorders) | 0 | 1
Pseudotumour - Operative Site (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Other - Operative Site (Infections and infestations) | 1 | 0 — Fever and red spot near wound
Other - Operative Site (Musculoskeletal and connective tissue disorders) | 1 | 0 — Migration of loose cerclage
Impingement - Operative Site (Musculoskeletal and connective tissue disorders) | 1 | 0
Other - Operative Site (Injury, poisoning and procedural complications) | 1 | 0 — Insufficient gluteus re-attachment
Operative Site - Other (Musculoskeletal and connective tissue disorders) | 0 | 1 — Swollen calf
Bronchopulmonary / Respiratory - Systemic (Respiratory, thoracic and mediastinal disorders) | 10 | 1
Carcinoma / Cancer - Systemic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 21 | 13
Cardiovascular - Systemic (Cardiac disorders) | 15 | 5
Cardiovascular - Systemic (Vascular disorders) | 1 | 0
Dermatological - Systemic (Skin and subcutaneous tissue disorders) | 1 | 1
Deep Vein Thrombosis (DVT) - Systemic (Vascular disorders) | 0 | 1
Gastrointestinal / Digestive - Systemic (Gastrointestinal disorders) | 7 | 6
Genitourinary / Urogenital - Systemic (Renal and urinary disorders) | 6 | 2
Musculoskeletal - Systemic (Musculoskeletal and connective tissue disorders) | 13 | 11
Musculoskeletal - Systemic (Nervous system disorders) | 0 | 1
Neurosensory / Neurological - Systemic (Nervous system disorders) | 9 | 5
Neurosensory / Neurological - Systemic (Vascular disorders) | 0 | 1
Pulmonary Embolism - Systemic (Vascular disorders) | 0 | 2
Thrombophlebitis - Systemic (Vascular disorders) | 1 | 0
Trauma - Systemic (Injury, poisoning and procedural complications) | 3 | 1
Death, Cause Unknown - Systemic (General disorders) | 3 | 3
Abdominal Pain - Systemic (Gastrointestinal disorders) | 0 | 2
Infection, Non-operative site - Systemic (Infections and infestations) | 0 | 3
Necrotizing Fascitis, Non-operative site - Systemic (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma, Non-operative site - Systemic (Musculoskeletal and connective tissue disorders) | 1 | 0
Epistaxis, Non-operative site - Systemic (Injury, poisoning and procedural complications) | 1 | 0
Wound Related, Non-operative site - Systemic (Injury, poisoning and procedural complications) | 0 | 1 — Complication associated with a wound from separate non-related surgery
Giant Cell Artheritis - Systemic (Vascular disorders) | 1 | 0
Bearing Wear, Non-operative Side - Systemic (Product Issues) | 1 | 0
Gynaecological - Systemic (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Accolade Stem (N=289) | Accolade II Stem (N=134)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 36 | 41

LIMITATIONS AND CAVEATS:
Registry-based study Modified HHS scores reported as unable to collect physical measurements in-person due to COVID-19 pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI may publish after study completion and prior multi-center publication, provided Sponsor reviews materials at least 15 working days before submission. Reasonable comments will be incorporated. Sponsor may request a delay of up to 1 month to protect proprietary information. For multi-center trials, site-specific publications cannot occur before the first multi-center publication unless otherwise agreed

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2013-08-30): https://cdn.clinicaltrials.gov/large-docs/44/NCT02520544/Prot_SAP_ICF_000.pdf